CLINICAL TRIAL: NCT02735356
Title: A Case Study of the Effects of Topical Itraconazole on Pharmacodynamic Modulation of Hedgehog Target Gene Expression in Basal Cell Carcinomas in Patients
Brief Title: Topical Itraconazole in Treating Patients With Basal Cell Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jean Yuh Tang (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jean Yuh Tang, Associate Professor of Dermatology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-35672; NCI-2016-00452 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SKIN0030 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Skin Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (itraconazole and placebo) (Experimental): Patients apply itraconazole topically BID and placebo topically BID for 12 weeks.
  Interventions: Drug: Itraconazole; Other: Placebo

INTERVENTIONS:
Drug: Itraconazole — Applied topically
  Other Names: Lozanoc; Oriconazole; R 51,211; Sporanox
Other: Placebo — Applied topically
  Other Names: placebo therapy; PLCB; sham therapy

SUMMARY:
This phase 0 trial studies how well itraconazole gel works in treating patients with basal cell cancer. Itraconazole gel may help to treat basal cell tumors in patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if 12 weeks of topical itraconazole gel reduces basal cell carcinoma (BCC) biomarkers (Gli1, the target gene of the Hedgehog pathway).

SECONDARY OBJECTIVES:

I. To determine if topical itraconazole gel will decrease BCC size.

OUTLINE:

Patients apply itraconazole topically twice daily (BID) and placebo topically BID for 12 weeks.

After completion of study treatment, patients are followed up for up to 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The subject must sign and date all informed consent statements; children will sign the assent form and their guardian will sign the consent form
* The subject must be willing to apply the medications twice daily for 1 month
* The subjects must have at least four BCCs in non-cosmetically sensitive sites
* For women of child-bearing potential, a negative urine pregnancy test
* Women of child-bearing potential are expected to use an effective method of birth control to prevent exposing a fetus to potentially dangerous agent with unknown risk
* For male patients with female partners of childbearing potential, agreement to use adequate contraception while you are participating in the study and 1 month after applying your last dose

Exclusion Criteria:

* Pregnancy or breast-feeding
* History of congestive heart failure or other findings of ventricular dysfunction
* History of current evidence of malabsorption or liver disease
* Current immunosuppression or taking immunosuppressive drugs
* Taking oral itraconazole
* Taking any medication known to affect hedgehog (HH) signaling pathway
* The subject has used topical or systemic therapies that might interfere with the evaluation of the study medication during the study; specifically these include the topical use to the study tumors of: glucocorticoids (ii) retinoids (e.g., etretinate, isotretinoin, tazarotene, tretinoin, adapalene) systemically or topically (iii) alpha-hydroxy acids (e.g., glycolic acid, lactic acid) to more than 5% of the skin during the six months prior to study entry (iv) 5-fluorouracil or imiquimod; also - treatment with systemic chemotherapy or agents known to be inhibitors of HH signaling within 60 days to starting study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Percentage change of GLi levels in treated vs untreated tumors | Up to 1 month
  will be assessed as relative GLi1 mRNA expression

SECONDARY OUTCOMES:
Change in BCC tumor size | At baseline, 1, 4, and 12 weeks
  Analyzed based on tumor size change (longest diameter, Response Evaluation Criteria in Solid Tumors [RECIST] criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Oro, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford Cancer Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes